CLINICAL TRIAL: NCT06418802
Title: Clinical Series Study of the Effects of STN-DBS on Gait in Parkinson's Disease Based on Wearable Devices.
Brief Title: Study of the Effects of STN-DBS on Gait in Parkinson's Disease.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023YF062-02
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experiment 1: Experimental group 1 (Experimental): PD Patient's gait were followed up at 1 month,3 months,6 months, and 1 year after bilateral STN-DBS surgery.
  Interventions: Procedure: STN-DBS surgery
- Experiment 1: Comparator group 1 (Active Comparator): PD patient's gait with optimal medical therapy before bilateral STN-DBS surgery.
  Interventions: Procedure: STN-DBS surgery
- Experiment 2: Experimental group 2 (Experimental): PD patient's gait with a short pulse width (30s) with bilateral STN-DBS.
  Interventions: Device: pulse width
- Experiment 2: Comparator group 2 (Active Comparator): PD patient's gait with the conventional pulse width (60 s) with bilateral STN-DBS.
  Interventions: Device: pulse width
- Experiment 3: Experimental group 3 (Experimental): PD patient's gait with frequency parameters(60,100, and 130HZ) with bilateral STN-DBS.
  Interventions: Device: frequency
- Experiment 3: Comparator group 3 (Active Comparator): PD patient's gait with the conventional frequency parameters with bilateral STN-DBS.
  Interventions: Device: frequency

INTERVENTIONS:
Procedure: STN-DBS surgery — bilateral subthalamic nucleus deep brain stimulation surgery
  Arms: Experiment 1: Comparator group 1; Experiment 1: Experimental group 1
Device: pulse width — a short pulse width (30s)
  Arms: Experiment 2: Comparator group 2; Experiment 2: Experimental group 2
Device: frequency — frequency parameters of STN-DBS (60,100, and 130HZ)
  Arms: Experiment 3: Comparator group 3; Experiment 3: Experimental group 3

SUMMARY:
Objectives: Parkinson's disease (PD) is the second most common degenerative disease of the nervous system. Postural instability/gait disorder (PIGD) is one of the motor symptoms of Parkinson's disease, which affects the quality of life of patients with Parkinson's disease. At present, deep brain stimulation（DBS）can significantly improve tremor and bradykinesia, but whether deep brain stimulation is effective for gait disorders is still a controversial topic. In addition, the previous gait assessment mainly focused on scales or simple walking tests, and appropriate and effective evaluation methods are needed to evaluate the efficacy of intervention for gait disorders in PD patients. Therefore, in view of these problems, this study will use wearable devices and traditional scale evaluation to explore the effects of deep brain stimulation on gait in patients with Parkinson's disease.

Methods: A total of 30 patients with Subthalamic nucleus DBS（STN-DBS）were expected to be enrolled. By adjusting the parameters of STN-DBS (voltage, frequency, pulse width), the effects of different parameters on PD gait were compared. Gait changes were mainly analyzed by wearable devices and MDS Unified Parkinson's Disease Rating Scale assessment（MDS-UPDRS）. The （Timed Up and Go）TUG test, narrow channel task, circle task and trajectory analysis were performed in the unmedicated state. The wearable device was used to collect the motion information of 10 different positions of the human body, including the wrist, thigh, ankle, foot tip, chest and waist nodes. (1)Experiment 1: Patients were divided into pre-operation group and post-operation group. A case-control study was conducted, and patients were followed up at 1 month,3 months,6 months and 1 year after operation. (2)Experiment 2: This study was a single-center, randomized, double-blind, crossover trial of deep brain stimulation with a short pulse width (30s) versus conventional pulse width (60 s) in PD patients with bilateral STN-DBS. Gait data and MDS-UPDRS were collected at baseline, after 4 weeks and 8 weeks. (3)Experiment 3: By adjusting the frequency parameters of STN-DBS (30,100, and 130HZ), gait data and MDS-UPDRS were collected after 10 minutes of the washout period, and the best DBS parameters for gait improvement were maintained for 4-8 weeks and then evaluated again.

Expected results: By adjusting the parameters (voltage, frequency, and pulse width) of STN-DBS, the potential mechanisms for improving gait disorders in PD were explored, meaningful digital biomarkers for PD gait prognosis were explored, and long-term programming of STN-DBS was guided.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 40-75 years old; (2) Patients who meet the Chinese Parkinson's disease diagnostic criteria and confirmed by two high-level physicians (>10 years); (3) Diagnosed by Parkinson's Specialty Clinic For Parkinson's disease for more than 1 year and have been effective after treatment; (4) Hearing, visual and cognitive abilities are normal; (5) The subjects were informed of the test purpose, the benefits of the test, the test process and possible unexpected situations before the test , and signed the trial informed consent form.

Exclusion Criteria:

* (1) A variety of secondary Parkinson's syndrome (including traumatic, drug-induced, tumor, vascular, toxic, hydrocephalus, etc.) and Parkinson's superimposed syndrome. (2) Other diseases that cause gait disorders, including spinal joint injuries, muscle spasm, stroke, peripheral neuropathy, muscle diseases, hydrocephalus, cognitive impairment, etc. (3) Accompanied by vital organ (heart, lung, liver, kidney, etc.) failure, malignant tumors, unstable conditions and other serious medical diseases. (4) Those who have serious behavior problems or mental confusion. (5)Those who do not cooperate with the examination.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Gait data | Pre-operation（baseline)，1 month,3 months,6 months and 1 year after operation.
  Gait changes were analyzed by wearable devices and MDS-UPDRS.
Gait data | Baseline, after 4 weeks and 8 weeks.
  Gait changes were analyzed by wearable devices and MDS-UPDRS.
Gait data | Baseline, after 10 minutes of the washout period, after4-8 weeks.
  Gait changes were analyzed by wearable devices and MDS-UPDRS.

IPD SHARING:
Plan to Share IPD: No